CLINICAL TRIAL: NCT03957486
Title: Effect of Arterial Cannulation on the Continuous and Non-invasive Hemoglobin Monitoring for Laparoscopic Gastrectomy
Brief Title: Effect of Arterial Cannulation on the Continuous and Non-invasive Hemoglobin Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Eun Kim, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AJIRB-MED-OBS-18-48
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Same group (Experimental): arterial cannulation on same arm of continuous hemoglobin monitoring
  Interventions: Other: arterila cannulation on same arm
- Different group (Placebo Comparator): arterial cannulation on different arm of continuous hemoglobin monitoring
  Interventions: Other: arterila cannulation on different arm

INTERVENTIONS:
Other: arterila cannulation on same arm — arterila cannulation on same arm receiving continous hemoglobin monitoring
  Arms: Same group
Other: arterila cannulation on different arm — arterila cannulation different arm receiving continous hemoglobin monitoring
  Arms: Different group

SUMMARY:
The primary purpose of this study is to investigate the effect of arterial cannulation on the continuous and non-invasive hemoglobin monitoring during laparoscopic gastrectomy

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic gastrectomy under general anesthesia

Exclusion Criteria:

* atypical hemoglobin disease, infective state, cardiovascular disease, peripheral vascular disease

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
difference between SpHb value and SaHb value (SpHb - SaHb) in g/dL | 3 time points from the start of anesthesia to the end of anesthesia, an average 2 hours
  SpHb value (g/dL) is measured by co-oxymetry, and SaHb value (g/dL) is measured by blood sampling.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Ajou University School of Medicine, Suwon, South Korea